CLINICAL TRIAL: NCT06514469
Title: Safety and Efficacy of Sufentanil Administration by Paramedics in Acute Trauma in Prehospital Setting: Observational Study
Brief Title: Safety and Efficacy of Sufentanil Administration by Paramedics in Acute Trauma
Status: Recruiting | Type: Observational
Sponsor: Zdravotnicka Zachranna Sluzba Karlovarskeho Kraje, P.O. (Other)
Responsible Party: Principal Investigator, Roman Sýkora, MD, Ph.D., Researcher, physician, Zdravotnicka Zachranna Sluzba Karlovarskeho Kraje, P.O.
Other Study IDs: Sufentanil02
Record Dates: First submitted 2024-07-16; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Injury Traumatic; Pain, Acute
Keywords: sufentanil; acute trauma; pain; paramedic; competence; prehospital
MeSH Terms: conditions — Wounds and Injuries; Acute Pain; Pain | interventions — Referral and Consultation; Mental Competency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Consultation: Patient who were administered sufentanil in acute trauma by paramedics after phone call consultation with medical doctor.
  Interventions: Drug: Sufentanil intravenous administration followed consultation of remote physician
- Competency: Patient who were administered sufentanil in acute trauma by paramedics based on their competencies.
  Interventions: Drug: Sufentanil intravenous administration based on paramedic competency

INTERVENTIONS:
Drug: Sufentanil intravenous administration followed consultation of remote physician — Intravenous administration of sufentanil to patients with acute injury by paramedics only after phone-call consultation of medical doctor.
  Other Names: Consultation
  Groups: Consultation
Drug: Sufentanil intravenous administration based on paramedic competency — Intravenous administration of sufentanil to patients with acute injury by paramedics based on their competencies
  Other Names: Competency
  Groups: Competency

SUMMARY:
The safety and efficacy of competence of paramedics to administer sufentanil intravenously in adult acute trauma patients without presence or without phone-call consult with an emergency medical doctor will be assessed in this observational study.

Condition or disease: pain in trauma or injury. Intervention/treatment: sufentanil administered by paramedics after the phone call consultation of medical doctor versus sufentanil administered by paramedics based on their competency, without consultation of medical doctor.

DETAILED DESCRIPTION:
The administration and indication of an opioid analgesics is carried by a medical doctor in most European emergency services. However, trips to majority of less serious traumas are realized by ambulances with paramedic crews without a medical doctor present on site.

This study will assess the new competence of paramedics to administer opioid analgesics without presence or phone-call consult with an emergency medical doctor.

This study will address the safety and efficacy of sufentanil administered by the paramedics in the field to patients with acute trauma without any consultation with medical doctors.

This study will complement the recently published data of the previous study, which, however, took place during the outbreak of COVID-19 and this lockdown situation could have distorted the frequency and nature of the observed cases.

ELIGIBILITY:
Inclusion Criteria:

* acute trauma with severe pain (VAS/NRS > 4)
* age > 18 years
* conscious patient (GCS = 15; alert in AVPU)
* haemodynamically stable patient (> 100mmHg of systolic blood pressure, > 60/min of heart rate)

Exclusion Criteria:

* EMS doctor on site
* paediatric patient (less than 18 years)
* predominantly chronic but not acute pain
* incomplete documentation
* other than traumatic reasons for opioid administration (eg. acute coronary syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prehospital emergency care Adults patient Acute trauma with severe pain.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
The safety of pain treatment by the paramedics with competence to sufentanil - administration in acute trauma - incidence of apnea | After sufentanil administration up to the handover of the patient to the hospital, up to 60 minutes.
  Measurement of incidence of adverse effects of sufentanil administration in both study groups - apnea - during the period from sufentanil administration (baseline) up to handover of the patient to the hospital (percentage).
The safety of pain treatment by the paramedics with competence to sufentanil - administration in acute trauma - incidence of bradypnoea | After sufentanil administration up to the handover of the patient to the hospital, up to 60 minutes.
  Measurement of incidence of adverse effects of sufentanil administration in both study groups - bradypnoea - is measured during the period from sufentanil administration (baseline) up to handover of the patient to the hospital (percentage).
The safety of pain treatment by the paramedics with competence to sufentanil - administration in acute trauma - incidence of nausea. | After sufentanil administration up to the handover of the patient to the hospital, up to 60 minutes.
  Measurement of incidence of adverse effects of sufentanil administration in both study groups - nausea - is measured during the period from sufentanil administration (baseline) up to handover of the patient to the hospital (percentage).
The safety of pain treatment by the paramedics with competence to sufentanil administration in acute trauma - incidence of vomiting | After sufentanil administration up to the handover of the patient to the hospital, up to 60 minutes.
  Measurement of incidence of adverse effects of sufentanil administration in both study groups - vomiting - is measured during the period from sufentanil administration (baseline) up to handover of the patient to the hospital (percentage).
The efficacy of pain treatment by the paramedics with competence to sufentanil - administration in acute trauma - NRS (numeric rating scale). | Before sufentanil administration and at the handover of the patient to the hospital, up to 60 minutes.
  The ten point Numeric rating scale is used to measure the efficacy of pain treatment. The difference of VAS before administration of sufentanil and at the handover at the emergency department is calculated and compared in both groups (in points).
The efficacy of pain treatment by the paramedics with competence to sufentanil - administration in acute trauma - visual analogue scale. | Before sufentanil administration and at the handover of the patient to the hospital, up to 60 minutes.
  The ten point Visual analogue scale is used to measure the efficacy of pain treatment. The difference of VAS before administration of sufentanil and at the handover at the emergency department is calculated and compared in both groups (in points).

SECONDARY OUTCOMES:
Dose of administered sufentanil | After sufentanil administration, up to 60 minutes
  The average dose of administered sufentanil per each case (in micrograms) is reported in both groups.
Incidence of potentiation of analgesia by other analgesics | After sufentanil administration, up to 60 minutes.
  Number of cases of potentiation of analgesia by use of additional analgesics and is reported and compared in both groups (pertcentage).
Types of drugs used for potentiation of analgesia by sufentanil | After sufentanil administration, up to 60 minutes.
  The type and generic name of additional analgesics and is reported and compared in both groups (pertcentage).
The influence on haemodynamic parameters - non invasive blood pressure (BP) -systolic blood pressure | Before sufentanil administration and at the time of the handover in hospital, up to 60 minutes.
  The difference of systolic blood pressure before the administration of sufentanil and at the handover at the emergency department is measured, calculated and compared in both groups. Systolic blood pressure is measured in milimeters of hydrargyrum (mmHg).
The influence on haemodynamic parameters - non invasive blood pressure (BP) - diastolic blood pressure | Before sufentanil administration and at the time of the handover in hospital, up to 60 minutes.
  The difference of diastolic blood pressure before the administration of sufentanil and at the handover at the emergency department is measured, calculated and compared in both groups. Diastolic blood pressure is measured in milimeters of hydrargyrum (mmHg).
The influence on haemodynamic parameters - heart rate (HR) | Before sufentanil administration and at the time of the handover in hospital, up to 60 minutes.
  The difference of heart rate before the administration of sufentanil and at the handover at the emergency department is measured, calculated and compared in both groups. Heart rate is measured as monitored or palpated beats per minute (bpm).
The influence on peripheral oxygen saturation (SpO2) | Before sufentanil administration and at the time of the handover in hospital, up to 60 minutes.
  The difference of SpO2 before the administration of sufentanil and at the handover at the emergency department is measured, calculated and compared in both groups. SpO2 is measured as percentage.
Need for oxygenotherapy | After sufentanil administration up to the handover of the patient to the hospital, up to 60 minutes.
  Measurement of incidence of need for oxygenotherapy is measured during the period from sufentanil administration (baseline) up to handover of the patient to the hospital (percentage).
Antiemetics usage | After sufentanil administration up to the handover of the patient to the hospital, up to 60 minutes.
  Antiemetic drugs used after sufentanil administration to treat nausea or vomiting (percentage).
Atropine usage | After sufentanil administration up to the handover of the patient to the hospital, up to 60 minutes.
  Atropin usage due to bradycardia after sufentanil administration (percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Jiří Smetana, MD, Study Director — Zdravotnická záchranná služba Karlovarského kraje, příspěvková organizace
Locations (1):
- Zdravotnická záchranná služba Karlovarského kraje, příspěvková organizace, Karlovy Vary, Karlovy Vary Region, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available upon request.

REFERENCES:
- [Result] Renza M, Sykora R, Peran D, Hricova K, Brizgalova N, Bakurova P, Kukacka M. Pilot implementation of the competence of Czech paramedics to administer sufentanil for the treatment of pain in acute trauma without consulting a physician: observational study. BMC Emerg Med. 2022 Apr 9;22(1):63. doi: 10.1186/s12873-022-00622-8. PMID 35397498
- [Result] Scharonow M, Alberding T, Oltmanns W, Weilbach C. Project for the introduction of prehospital analgesia with fentanyl and morphine administered by specially trained paramedics in a rural service area in Germany. J Pain Res. 2017 Nov 6;10:2595-2599. doi: 10.2147/JPR.S151077. eCollection 2017. PMID 29158691